CLINICAL TRIAL: NCT02459821
Title: The Effects of an Innovative Gait Robot for the Repetitive Practice of Floor Walking and Stair Climbing up and Down in Patients Suffered From Multiple Sclerosis: a Randomized Control Trial
Brief Title: Effects of GE-O System on Gait Impairments in Multiple Sclerosis Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Nicola Smania, MD, Clinical Professor, Prof. Nicola Smania, Universita di Verona
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GEO-SM2012JP
Record Dates: First submitted 2015-05-25; First posted 2015-06-02 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Gait rehabilitation; Quality of life; Stair climbing; Robotic
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Robot-assisted gait training group (Experimental): The first group will be subjected to RAGT for 9 weeks (2 sessions/ week) with a total of 18 sessions by mean of GE-O System (9). During each session, the patients will practice 15 to 20 min of simulated floor walking followed by 5 to 10 min of repetitive simulated stair climbing up and down. Breaks will be optional, but uninterrupted training intervals of at least 5 min for simulated floor walking and 3 min of simulated stair climbing will be required. When the patient reaches the maximum amount of time, speed of gait will then be progressively increased. Each session will last up to 50 minutes, the first 30 minutes will be dedicated to gait training and the last 20 minutes to stretch the lower limb's muscles.
  Interventions: Other: GE-O SYSTEM
- Conventional training group (Active Comparator): The group will be subjected to conventional gait training for 9 weeks (2 sessions/week) with a total of 18 sessions. Each session will last altogether 50 minutes, the first 30 minutes will be dedicated to gait and stair climbing up and down training while the last 20 minutes to stretch the lower limb's muscles.
  Interventions: Other: Conventional training

INTERVENTIONS:
Other: GE-O SYSTEM — The first group will be subjected to RAGT for 9 weeks (2 sessions/ week) with a total of 18 sessions by mean of GE-O System (9). During each session, the patients will practice 15 to 20 min of simulated floor walking followed by 5 to 10 min of repetitive simulated stair climbing up and down. Breaks will be optional, but uninterrupted training intervals of at least 5 min for simulated floor walking and 3 min of simulated stair climbing will be required. When the patient reaches the maximum amount of time, speed of gait will then be progressively increased. Each session will last up to 50 minutes, the first 30 minutes will be dedicated to gait training and the last 20 minutes to stretch the lower limb's muscles.
  Arms: Robot-assisted gait training group
Other: Conventional training — The conventional walking group will be subjected to a conventional gait training for 9 weeks (2 sessions/week) with a total of 18 sessions. Each session will last altogether 50 minutes, the first 30 minutes will be dedicated to gait and stair climbing up and down training while the last 20 minutes to stretch the lower limb's muscles.
  Arms: Conventional training group

SUMMARY:
Multiple sclerosis (MS) is the most common non-traumatic cause of neurologic disability in young adults,affecting mobility and ambulation in the majority of patients. At least 50% of individuals with MS will require an assistive device to ambulate within ten years of diagnosis. Impaired mobility is one of the top three factors associated with inability to continue working. In addition,impaired mobility and the inability to walk functionally translate into significant costs for personal assistance, medical complications, and lost wages because of unemployment. Clearly,maximizing the ability to ambulate, as well as perform safe and effective transfers,is a fundamental goal in the management of individuals with MS. None of the currently available MS disease-modifying medications have been shown to stop or reverse gait disability. Repetitive locomotor training is an innovative approach in gait disturbances in patients with MS. Only scant data on this issue is available and all the studies have been performed by means of treadmill training or robot assisted gait training (RAGT) approaches. The recent introduction of a robotic device to gait rehabilitation showed a significant improvement in gait ability in patients with neurological disease due to the possibility of being trained under a graduated body weight support condition and being being guided to reproduce a physiologic gait pattern.

In 2010 a novel device called GE-O System was developed. It enables patients to repetitively practice walking on the floor and also climb up and down stairs. To date, the effectiveness of this novel device has not yet been evaluated in patients with MS. The aims of the study are as follows: to evaluate the effectiveness of a specific gait training program consisting of the GE-O System in patients with MS in improving balance and walking ability,reducing fatigue,the frequency of falls,the fear of falling and disability in activities of daily living and finally,improving quality of life.

DETAILED DESCRIPTION:
Material and methods Stages of the study and deadlines

1. Presentation of the study to collaborating unit: 1 months
2. Patient recruitment and evaluation: 3 months
3. Assessment and treatment procedures: 9 months
4. Follow-up evaluation: 10 months
5. Data analysis: 1 year

   STAGE A. PRESENTATION OF THE STUDY

   The first stage of the program consists of:
   1. Conduct meetings between the operators of the Neurological and Cognitive Rehabilitation Research Centre, Department of Neurological, Neuropsychological, Morphological and Movement Sciences of the University of Verona, and Neurological Unit of Policlinic Hospital, Verona, Italy
   2. Train all collaborating medical doctors and physical therapists with regards to the purposes of the study, patient recruitment protocol, treatment methodology and data collection procedures.

   STAGE B. RECRUITMENT AND EVALUATION
   1. All the patients with MS referred to the above mentioned Unit over the first 3 months of the study will be examined;
   2. Medical doctors operating in these units will fill out a data collection card for each patient;
   3. Patients meeting the inclusion criteria will be recruited;
   4. Medical doctors of the Units will refer the selected patients to the main investigator;
   5. Informed consent for participating in the study will be obtained;
   6. Patients recruited will be evaluated by means of clinical and instrumental procedures
   7. Before treatment evaluation (T0): 6-Minute Walking Test, 10-Metre Walking Test, Berg Balance Scale, Activities-specific Balance Confidence Scale, Fatigue Severity Scale, Stair Climbing Test, Multiple Sclerosis Quality Of Life-54, gait analysis, electromyography and stabilometric assessments.

   STAGE C. ASSESSMENT AND TREATMENT PROCEDURES
   1. Patients will be assigned to 2 groups, matching on sex, age, severity of disease and primary outcome measure (6MWT). The Principal Investigator will hold the list of patients.
   2. Patients allocated in the Group 1 will perform robot-assisted gait training by means of GE-O System. Patients allocated in the Group 2 will perform conventional walking rehabilitation.
   3. After treatment evaluation (T1): the clinical and instrumental procedures applied at T0 will be repeated at the end of treatment.

   STAGE D. FOLLOW-UP EVALUATION
   1. Follow-up evaluation (T2): the clinical and instrumental procedures applied at T0 and T1 will be repeated 1 month post-treatment.

      STAGE E. DATA ANALYSIS All data collected from the patients will be examined. The data will then be transferred into electronic sheets and processed with statistics programs.

      Subjects The study will include 48 (see statistical section) patients with definite diagnosis of MS, as determined clinically (8).

      Inclusion Criteria will be:

      • Expanded Disability Status Scale (EDSS) between 3 and 6.5;
      * Mini Mental Examination State >24;
      * Absence of cognitive impairment;
      * Age <75 years;
      * Absence of heart failure;
      * Ability to sit without trunk support;
      * Ability to stand for at least 10 seconds with support;
      * Absence of concurrent neurological or orthopaedic diseases that interfere with deambulation;

      Exclusion criteria:

      • Those patients with disease recurence that worsens significantly during the 8 weeks before recruitment;
      * changes in pharmacological therapy that could modified disease course in the previous three months;
      * changes in pharmacological therapy for fatigue treatment in the previous three months;
      * performance of any type of rehabilitation treatment in the month prior to recruitment.

      Study plan It is a controlled randomised clinical trial, with blinded assessments in two groups of patients with MS. The allocation in the groups will be done with simple randomisation scheme (www.randomization.com).

      Group 1 - Robot-assisted gait training The first group will be subjected to RAGT for 6 weeks (2 sessions/ week) with a total of 12 sessions by mean of GE-O System (9). During each session, the patients will practice 15 to 20 min of simulated floor walking followed by 5 to 10 min of repetitive simulated stair climbing up and down. Breaks will be optional, but uninterrupted training intervals of at least 5 min for simulated floor walking and 3 min of simulated stair climbing will be required. When the patient reaches the maximum amount of time, speed of gait will then be progressively increased. Each session will last up to 50 minutes, the first 30 minutes will be dedicated to gait training and the last 20 minutes to stretch the lower limb's muscles.

      Device - GE-O System ("Rehatecnologies" Company, "Bozen", Italy) The device follows the end effector principle. The harness secured patient stood on two foot plates, whose trajectories are completely programmable. The two foot plates are connected each by a pivoting arm to two moving sledges. The foot's forward motion is given by the movement of the principal sledge, which is connected to the transmission belt of the linear guide. The transmission belt is driven by a 1.500 W servomotor fixes to the back end of the linear guide. The forward and backward excursion of the principal sledge ensure the control of the step length. The mechanic design for the control of the step height is realized implementing the scissor principle. The second sledge on the linear guide moves relatively to the principal sledge. A rod ensures the connection of the relative sledge to the pivoting arm. Nearing the relative sledge to the principal sledge closes the scissor, providing the pivoting arm to get lifted, and viceversa. The servomotor responsible for the relative motion is fixed under the relative sledge and connected to the principal sledge by a screw axle. A third completely programmable 400 W drive is fixed on the arm and transferred the rotation through a transmission belt to an external axle, which is aligned to the ankle, controlling the plantar- and dorsiflexion during the steps. The motion control of each servomotor is provided by an industrial personal computer, which is coupled to the eight motion controllers responsible for each programmable degree of freedom on the machine, three for each leg and two for the CoM control. The maximal step length corresponds to 55 cm, the maximal achievable angles were ± 90°. The step height in the workspace is 40 cm, allowing the patient to climb a standardized step of 18 cm. The maximal possible gait velocity is 0,6 m/s. The feet are placed in two snowshoe bindings on a steel plate, which was fixed to the basis plate by magnets. The plate looseness in all three directions of the footplate, if a limit momentum of 4 Nm was exceeded. Hand rails at both sides are settable vertically and laterally. The patient's body weight support system is fixed by an aluminium chassis. It consisted of an electrical patient lift system, intends for helping the patients to stand up from the wheelchair, and a drive activating a three roll mechanism. The patent lifter's belt passes through the three rolls mechanism and is attached to patient's harness. The belt got shorten by the mechanism's motion, ensuring the vertical motion of patient's centre of mass (CoM). The two ends of a rope are fixed to patient's harness at hip height to control the lateral motion of patient's CoM. Another drive moves the rope. A ramp allows wheelchair access into the device from behind, to be followed by getting in the snowshoes, fastening them, securing the patient lifter's belt to the harness, standing up with the assistance of the therapist, and a last check before starting therapy. The graphic user interface (GUI) showed the actual trajectories for any of the conditions on-line, so that the therapist will be able to control and to correct it. Changes could be made for step length, step height, the toe off and the initial contact inclination angles of the feet. For a perfect match of the listed trajectory settings, the patient will be fixed in the snowshoe bindings in such a way that the marked position of the metatarsale V in the binding corresponded to the patient's metatarsale V. The therapist could further adapt the excursions of the CoM in the vertical and horizontal directions and the relative position of the suspension point with respect to the footplates. The PC memorizes the treatment conditions of each individual patient. The dimensions of the CE-certified machine (medical device directive 93/42/EEC) are 2.800 mm 1.200 mm 2.300 mm, the net weight was 850 kg, the power supply was 230 V.

      Group 2 - Conventional walking group (CW) The CW group will be subjected to conventional gait training for 6 weeks (2 sessions/week) with a total of 12 sessions. Each session will last altogether 50 minutes, the first 30 minutes will be dedicated to gait and stair climbing up and down training while the last 20 minutes to stretch the lower limb's muscles.

      Assessment procedures All of the patients enlisted at every evaluation will undergo the following clinical and instrumental evaluations by the same physician unaware to the treatment allocation.

      Clinical assessments:

      • 6-Minute Walking Test: this is a validated tool evaluating walking capacity. Subjects will be required to walk at their maximum speed for 6 minutes and the score will be the covered distance (10).

      • 10-Metre Walking Test: this test has been selected as a measure of gait speed. This is a validated test requiring to walk on a flat hard floor at patient's fastest speed for 10 metres. Scoring will be walking speed (11).

      • Berg Balance Scale: this is a performance-based assessment tool used to evaluate standing balance during functional activities. This scale rates performance from 0 (cannot perform) to 4 (normal performance) on 14 items (corresponding to 14 tasks such as sitting, changing position, transferring, standing, turning, stepping and reaching) with a maximum total score of 56 (12).

      • Activities-specific Balance Confidence Scale: this is a scale in which the subject rates his or her perceived level of confidence while performing 16 daily living activities (such as walking, bending, standing and reaching) (13).

      • Fatigue Severity Scale: This is a validated scale used to assess fatigue. It consists of a self-report questionnaire composed of 9 items. Each item is scored from 1 (absence of fatigue) to 7 (high level of fatigue). The score ranges from 9 to 63 (14).

      • Stair Climbing Test: the test will be performed as a symptom limited exercise. The patients will be asked to climb, at a pace of their own choice, the maximum number of steps and to stop only for exhaustion, limiting dyspnea, leg fatigue, or chest pain. During the exercise, pulse rate and capillary oxygen saturation will be monitored by means of a portable pulse oximeter (15).

      • Multiple Sclerosis Quality Of Life-54: This is a validated multidimensional health-related quality of life measure. This 54-item instrument generates 12 subscales along with 2 summary scores, and 2 additional single-item measures. The summary scores are the physical and mental health composite summaries (16).

      Instrumental assessment procedures
      * Gait Analysis: It is an electronic system used for the gathering of the temporal-spatial data of deambulation. It is made up of an 8 meter long walkway connected to a PC. The system records the signal, reproducing the pressure maps of each step on video, identifying the progression of the center of gravity and recording all of the temporal-spatial features of gait (17).
      * Electromyographic analysis: the electromyographic activity of seven lower limb muscles of the both side (Mm. tibialis anterior, gastrocnemius, vastus medialis, vastus lateralis, rectus femorals, biceps femorals, and gluteus medius) will be detected by pairs of self-adhesive surface electrodes (diameter 8 mm) following a standardized protocol: the electrodes will be attached 2 cm apart on the muscle bellies after a conventional skin preparation (shaving, cleansing, and abrasion of keratinized epidermis). The impedance will be checked and keep below 5 kΩ. Signals (sampling rate 1.000 Hz) will be pre-amplified with standard preamplifiers of the system attached to the limb and memorize by the portable data logger (9).
      * Stabilometric assessment: the static balance will be carried out with a monaxial platform, an electronic system used for the evaluation of the instant position of the centre of pressure (CoP), the calculation of the anterior-posterior (AP)/medial-lateral (ML) body sway, the length of CoP trajectory and the speed of AP and ML CoP displacements. It is made up of a square dynamometric platform connected to a PC (18)

      Criteria of interruption of the treatment and withdrawal from the study.

      The patient at any moment may drop out of the study. Furthermore, it is necessary to suspend treatment and withdraw from the study if:
      * Cardio-Respiratory complications arise that may or may not depend on the exercise.
      * Any other condition that may alter the patient's general health even if it does not depend on the treatment.

      Ethical aspects The study will be submitted to the local ethical committee. The data gathered during this study will be available and accessible only to the personnel involved, to the ethical committee and to the Ministry for Health, as stated by local laws (L. 675/96).

      Statistical elaboration A prestudy power calculation estimated to enrol at least 48 subjects providing 90% power to detect a clinical significant difference in the 6MWT of 55 meters between the 2 groups. Sample characteristics will be summarised using descriptive statistics, means, standard deviations, range and median values. Parametric and nonparametric tests will be performed according to variable distribution (19). Differences between and within groups at T0, T1 and T2 will tested using Anova or Kruskal Wallis test. Differences between and within groups at T0, T1 and T2 as well as the correlation between outcomes will be tested. The alpha level will be set for significance at 0.05, however, to adjust for multiple comparison the "Bonferroni" correction will be used (alpha=0.025). Data will be analysed using SPSS software (version 16.0; SPSS Inc., Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* Expanded Disability Status Scale (EDSS) between 3 and 6.5;
* Mini Mental Examination State >24;
* Absence of cognitive impairment;
* Age <75 years;
* Absence of heart failure;
* Ability to sit without trunk support;
* Ability to stand for at least 10 seconds with support;
* Absence of concurrent neurological or orthopaedic diseases that interfere with deambulation;

Exclusion Criteria:

* Those patients with disease reccurence that worsens significantly during the 8 weeks before recruitment;
* changes in pharmacological therapy that could modified disease course in the previous three months;
* changes in pharmacological therapy for fatigue treatment in the previous three months;
* performance of any type of rehabilitation treatment in the month prior to recruitment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-05; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
6-Minute Walking Test (meters) | All patients enrolled in the study will be evaluated before the beginning (baseline time 0) of treatment and after the end (after 6 weeks) of the treatment.
  Change from Baseline in meters at 6 weeks

SECONDARY OUTCOMES:
10-Metre Walking Test (seconds) | All patients enrolled in the study will be evaluated before the beginning (baseline time 0) of treatment and after the end (after 6 weeks) of the treatment.
  Change from Baseline in seconds at 6 weeks
Berg Balance Scale | All patients enrolled in the study will be evaluated before the beginning (baseline time 0) of treatment and after the end (after 6 weeks) of the treatment.
  Change from Baseline in score at 6 weeks
Activities-specific Balance Confidence Scale | All patients enrolled in the study will be evaluated before the beginning (baseline time 0) of treatment and after the end (after 6 weeks) of the treatment.
  Change from Baseline in score at 6 weeks
Fatigue Severity Scale | All patients enrolled in the study will be evaluated before the beginning (baseline time 0) of treatment and after the end (after 6 weeks) of the treatment.
  Change from Baseline in score at 6 weeks
Stair Climbing Test (seconds) | All patients enrolled in the study will be evaluated before the beginning (baseline time 0) of treatment and after the end (after 6 weeks) of the treatment.
  Change from Baseline in seconds at 6 weeks
Multiple Sclerosis Quality Of Life-54 | All patients enrolled in the study will be evaluated before the beginning (baseline time 0) of treatment and after the end (after 6 weeks) of the treatment.
  Change from Baseline in score at 6 weeks
Gait Analysis | All patients enrolled in the study will be evaluated before the beginning (baseline time 0) of treatment and after the end (after 6 weeks) of the treatment.
  Change from Baseline in spatiotemporal gait parameters at 6 weeks
Stabilometric assessment | All patients enrolled in the study will be evaluated before the beginning (baseline time 0) of treatment and after the end (after 6 weeks) of the treatment.
  Change from Baseline in stabilometric score at 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Smania, MD, Principal Investigator — Neuromotor and Cognitive Rehabilitation Center Department of Neurological and Movement Sciences University of Verona, Verona, Italy P.zza L.A. Scuro, 10 37134 Verona, Italia
Locations (2):
- Italy (2):
  - Azienta Ospedaliera, SSO Rehabilitation Unit, Verona, Verona, Italy, Verona
  - prof. Smania Nicola, Verona, Verona